CLINICAL TRIAL: NCT00792259
Title: Topcon 3D OCT-1000 Optical Coherence Tomography System for Measurements of Retinal and RNFL Thicknesses: Precision and Agreement Study
Brief Title: Topcon 3D OCT-1000 Optical Coherence Tomography System
Status: Completed | Type: Observational
Sponsor: Topcon Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Organization: Topcon Corporation (Industry)
Other Study IDs: Topcon 01
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Results first posted 2015-06-17 (Estimated); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Retinal Disease; Glaucoma
MeSH Terms: conditions — Retinal Diseases; Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Patients with Retinal Disease
- 2: Patients without Retinal Disease
- 3: Normal Subjects

SUMMARY:
The purpose of this clinical protocol is to perform a comparison of Retinal and Retinal Nerve Fiber Layer (RNFL) thickness measurements between the Topcon 3D-1000 and the identified predicate device. In addition, this protocol performs a comparison of the thickness measurement results from images collected and analyzed with the Zeiss Stratus OCT to images collected with the Zeiss Stratus OCT and imported into the Topcon 3D OCT-1000 StratusViewer for analysis.

ELIGIBILITY:
Retinal Disease Study

No Retinal Disease:

Inclusion Criteria:

* Male or female
* Between 18 and 80 years of age
* Either eye, but only one eye per subject will be enrolled
* Topcon image quality factor ≥ 45 or Stratus signal strength ≥ 5.

Exclusion Criteria:

* Any known ocular disease
* Any systemic disease that could result in ocular manifestations such as hypertension, diabetes, heart disease, etc.
* Topcon image quality factor ≤ 44 or Stratus signal strength < 5.

Retinal Disease

Inclusion Criteria:

* Male or female
* Between 18 and 80 years of age
* Either eye, but only one eye per subject will be enrolled
* Symptoms consistent with one of the following retinal diseases: diabetic macular edema, cystoid macular edema, epiretinal membrane, macular hole, wet AMD and dry AMD for which OCT imaging is warranted. At lease one (1) case each of these diseases will be included in the study
* A range of retinal thickness will be included
* Topcon image quality factor ≥ 45 or Stratus signal strength ≥ 5.

Exclusion Criteria:

* Presence of glaucoma
* Topcon image quality factor ≤ 44 or Stratus signal strength < 5.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ophthalmology practice
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2008-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Retina Consultations, Bronxville, New York
  - New York Eye and Ear-Glaucoma Associates of New York, New York, New York
  - Vitreous-Retina-Macula Consultants of NY, New York, New York
  - SUNY, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Retinal Disease Eyes: Retinal Disease subjects with ocular pathology
- Normal Subjects: Normal subjects with no known ocular pathology
- Glaucoma Subjects: Subjects presented with Glaucoma
Period: Overall Study
Arm/Group | Retinal Disease Eyes | Normal Subjects | Glaucoma Subjects
Started | 15 | 20 | 13
Completed | 14 | 20 | 13
Not Completed | 1 | 0 | 0
Not completed — Poor Quality Scans | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 20 Normal Subjects 15 Retinal Disease subjects 13 Glaucoma Subjects
Groups:
- Retinal Disease Subjects: Retinal Disease subjects with ocular pathology
- Glaucoma Subjects: Glaucoma subjects presented with pathology
- Total: Total of all reporting groups
Arm/Group | Normal Subjects | Retinal Disease Subjects | Glaucoma Subjects | Total
Number analyzed (Participants) | 20 | 15 | 13 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 5 | 9 | 34
  >=65 years | 0 | 10 | 4 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.45 (10.36) | 66.6 (13.92) | 59.1 (17.63) | 50.52 (20.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 9 | 33
  Male | 6 | 5 | 4 | 15
Region of Enrollment [Number; unit: participants]
  United States | 20 | 15 | 13 | 48

OUTCOME MEASURES:

1. Primary Outcome: Precision and Agreement Between the Topcon 3D OCT 1000 and the Identified Predicate Device
Description: The precision and agreement measures the thickness of RNFL and Full Retinal Thickness of the study device and is compared to the predicate device to show agreement.
  Keywords, ILM - Internal Limiting Membrane RPE - Retinal Pigment Epithelium RNFL - Retinal Nerve Fiber Layer
Time Frame: 30 Minutes
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Normal Subjects | Retinal Disease Eyes | Glaucoma Subjects
Number analyzed (Participants) | 20 | 15 | 13
µm
  Retinal Thickness ILM-IS/OS 3D OCT-1000 | 235.0 (9.03) | 236.1 (48.06) | NA (NA) — Subject group not observed for this measurement
  Retinal Thickness ILM-IS/OS Stratus | 236.0 (12.54) | 263.1 (48.66) | NA (NA) — Subject group not observed for this measurement
  Retinal Thickness ILM-RPE 3D OCT-1000 | 252.8 (7.68) | 279.5 (45.36) | NA (NA) — Subject group not observed for this measurement
  Retinal Thickness ILM-BM 3D OCT-1000 | 296.0 (8.97) | 318.5 (41.90) | NA (NA) — Subject group not observed for this measurement
  RNFL Thickness 3D OCT-1000 | 107.4 (10.50) | NA (NA) — Subject group not observed for this measurement | 70.7 (19.87)
  RNFL Thickness Stratus | 105.9 (9.98) | NA (NA) — Subject group not observed for this measurement | 72.1 (20.25)

ADVERSE EVENTS:
Time Frame: 1 hour
Arm/Group | Retinal Disease Eyes | Normal Subjects | Glaucoma Subjects
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/20 | 0/13
Other Adverse Events (participants affected / at risk) | 0/15 | 0/20 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No